CLINICAL TRIAL: NCT02964598
Title: Sleep Helsinki! CIRCADIAN SLEEP REGULATION IN ADOLESCENCE
Brief Title: SleepHelsinki! CIRCADIAN SLEEP REGULATION IN ADOLESCENCE
Acronym: SleepHel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Helsinki (Other)
Collaborators: Academy of Finland (Other)
Responsible Party: Principal Investigator, Anu-Katriina Pesonen, Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1287174
Record Dates: First submitted 2016-11-09; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Sleep Disorder Circadian Rhythm, Delayed Sleep Phase Type
Keywords: Adolescent; Population-based; Social jetlag; Intervention; Bright light; Motivation; Circadian regulation; Behavioral change
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Control (Experimental): Minimal information on sleep timing
  Interventions: Other: Control
- Psychoeducation (Experimental): An extensive psychoeducational platform
  Interventions: Other: Psychoeducation
- Bright light (Experimental): Bright light treatment with 10 000 lux at max
  Interventions: Device: Bright light
- Gamified intervention (Experimental): A new gamified intervention designed for mobile phones
  Interventions: Behavioral: Gamified intervention
- Bright light and gamified intervention (Experimental): A combination of the two
  Interventions: Behavioral: Gamified intervention; Device: Bright light
- Sleep coaching (Experimental): A new intervention protocol including a personified approach to solve problems and increase motivation for better sleep behavior
  Interventions: Behavioral: Sleep coaching
- Sleep coaching + bright light (Experimental): A combination of the two
  Interventions: Behavioral: Sleep coaching; Device: Bright light

INTERVENTIONS:
Behavioral: Gamified intervention — A new mobile application for assisting in sleep regulation, duration 4-6 weeks
  Other Names: Helsinki Sleep Factory
  Arms: Bright light and gamified intervention; Gamified intervention
Behavioral: Sleep coaching — A new personalized program, duration 4-6 weeks
  Arms: Sleep coaching; Sleep coaching + bright light
Device: Bright light — Morning bright light 10 000 lux maximum duration 4-6 weeks
  Arms: Bright light; Bright light and gamified intervention; Sleep coaching + bright light
Other: Control — Minimal information on sleep timing and advancing the sleep rhythm
  Arms: Control
Other: Psychoeducation — An extensive information platform in the internet created for this purpose
  Arms: Psychoeducation

SUMMARY:
Adolescence associates with alterations in sleep-wake organization, such as later circadian phase preference. Simultaneously external pressures, such as evening-driven social activities increase. These may lead to delayed sleep phase, which may cause serious problems for waking up at socially accepted times, and absenteeism from the school may follow. This project aims at tracking risk factors for later circadian regulation problems, characterizing interconnections of biological, psychological and behavioural mechanisms that maintain or induce poor sleep regulation in adolescence, and building a cost-effective, theoretically-based sleep intervention for adolescents with delayed sleep phase. This randomized control trial capitalizes on a new population-based cohort of 16-17-year olds.

ELIGIBILITY:
Inclusion Criteria:

* Late bedtime several times per week

Exclusion Criteria:

* Chronic disease that affects sleep. Ongoing therapeutic treatment relationship if considered overlapping by the participant

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 270 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Circadian sleep rhythm | 8 weeks
  Actigraphy (brand GeneActiv)
Circadian body temperature rhythm | 8 weeks
  iButton measurement from the wrist

SECONDARY OUTCOMES:
Mood | 8 weeks
  Experience sampling method, brand Psymate
Insomnia symptoms | 8 weeks
  Bergen Insomnia Scale
Sleep problems | 8 weeks
  Pittsburgh Sleep Quality Index
Depression | 8 weeks
  Beck Depression Inventory
Anxiety | 8 weeks
  Generalized Anxiety Disorder questionnaire GAD-7

CONTACTS AND LOCATIONS:
Overall Officials: Anu-Katriina Pesonen, PhD, Principal Investigator — University of Helsinki
Locations (1):
- University of Helsinki, Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No